CLINICAL TRIAL: NCT06034626
Title: Therapeutic Effectiveness of Different Machines in Intense Pulsed Light Treatment of Meibomian Gland Dysfunction
Acronym: MGD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Aier Eye Hospital, Wuhan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-210
Record Dates: First submitted 2023-08-29; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: MGD-Meibomian Gland Dysfunction
Keywords: MGD; IPL; Non-inferiority analysis
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Intervention Model Description: The trial aimed to assess therapeutic effectiveness of the study treatment arm (OPL-I with the dual filter system; Miracle Laser systems, Wuhan, China) to the control treatment arm (M22 with a single filter; Lumenis, Yokneam, Israel). Each MGD patient underwent three treatment sessions at three-week intervals and three follow-up examinations over the course of treatment.
Who Masked: Participant
Masking Description: Patients receiving IPL treatment were masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPL-I (Experimental): Patients treated with OPL-I with the dual filter system
  Interventions: Procedure: Intense pulsed light; Drug: 0.3% hyaluronic acid eye drops
- M22 (Active Comparator): Patients treated with OPL-I with the single filter system
  Interventions: Procedure: Intense pulsed light; Drug: 0.3% hyaluronic acid eye drops

INTERVENTIONS:
Procedure: Intense pulsed light — Each MGD patient underwent three treatment sessions at three-week intervals and three follow-up examinations over the course of treatment.
Drug: 0.3% hyaluronic acid eye drops — 0.3% hyaluronic acid eye drops (Hialid; Santen, Osaka, Japan) four times a day during the study, including the follow-up period.

SUMMARY:
This study aimed to determine the therapeutic effectiveness of different machines in intense pulsed light (IPL) treatment of meibomian gland dysfunction (MGD). Subjects diagnosed with MGD underwent three sessions of IPL treatment in a control (M22) treatment group or experimental (OPL-I) treatment group and were followed up three to four weeks after each session. Tear breakup time (TBUT), meibomian gland secretion scores (MGSS), meibomian gland meibum scores (MGMS), corneal fluorescein staining (CFS) scores, and the Standard Patient Evaluation of Eye Dryness (SPEED) was used to assess eye dryness signs and symptoms at baseline and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Fitzpatrick skin type I-IV according to sun sensitivity and skin appearance
2. A Standard Patient Evaluation of Eye Dryness (SPEED) score of ≥6
3. Tear breakup time (TBUT) of ≤10 s in the studied eye
4. Corneal fluorescein staining (CFS) score of ≥1 (it is not necessary to consider this criterion if the TBUT is ≤5 s)
5. Meibomian gland secretion score (MGSS) of ≥6 in the studied eye.

Exclusion Criteria:

1. Use of prescription eye drops (excluding artificial tears) within 48 hours of recruitment
2. Facial IPL treatment within the prior 12 months
3. Any surgery of the eye or eyelids within the prior six months
4. Ocular surface and eyelid abnormalities
5. Any systemic condition that might cause eye dryness
6. Use of photosensitive drugs within the prior three months
7. Precancerous lesions
8. Skin cancer or pigmented lesions in the treatment area
9. Overexposure to the sun within the previous month
10. Ocular infections within the previous six months
11. Uncontrolled infections or immunosuppressive diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
SPEED Scores | Baseline, 1 month, 2 months, 3 months, 4 months
  Standard Patient Evaluation of Eye Dryness questionnaire
CFS scores | Baseline, 1 month, 2 months, 3 months, 4 months
  corneal fluorescein staining scores
TBUT | Baseline, 1 month, 2 months, 3 months, 4 months
  Tear breakup time
MGSS | Baseline, 1 month, 2 months, 3 months, 4 months
  Meibomian gland secretion scores. The MGSS evaluates the obstruction of meibum along the lower eyelid. Three positions along the lower eyelid were detected (five nasal, five central, and five temporal meibomian glands). A score of 0 indicated secretion by all five glands, a score of 1 indicated secretion by three to four glands, a score of 2 indicated secretion by one or two glands, and a score of 3 indicated no secretion by any glands.
MGMS | Baseline, 1 month, 2 months, 3 months, 4 months
  meibomian gland meibum scores. The MGMS evaluates the quality of meibum along the lower eyelid, with a score of 0 indicating clear liquid meibum, a score of 1 indicating cloudy liquid meibum, a score of 2 indicating cloudy granular meibum, and a score of 3 indicating toothpaste-like solid meibum).

SECONDARY OUTCOMES:
BCVA | Baseline, 4 months
  best-corrected visual acuity
IOP | Baseline, 4 months
  intraocular pressure measurements

CONTACTS AND LOCATIONS:
Overall Officials: Xiuming Jin, PhD, Study Director — Eye Center of the 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (3):
- China (3):
  - Hankou Aier Eye Hospital, Wuhan，Hubei Province, Wuhan, Hubei
  - Wuhan Aier Eye Hospital, Wuhan，Hubei Province, Wuhan, Hubei
  - 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
For patients' privacy reasons

REFERENCES:
- [Background] Toyos R, McGill W, Briscoe D. Intense pulsed light treatment for dry eye disease due to meibomian gland dysfunction; a 3-year retrospective study. Photomed Laser Surg. 2015 Jan;33(1):41-6. doi: 10.1089/pho.2014.3819. PMID 25594770
- [Background] Yan X, Hong J, Jin X, Chen W, Rong B, Feng Y, Huang X, Li J, Song W, Lin L, Cheng Y. The Efficacy of Intense Pulsed Light Combined With Meibomian Gland Expression for the Treatment of Dry Eye Disease Due to Meibomian Gland Dysfunction: A Multicenter, Randomized Controlled Trial. Eye Contact Lens. 2021 Jan 1;47(1):45-53. doi: 10.1097/ICL.0000000000000711. PMID 32452923